CLINICAL TRIAL: NCT00431743
Title: Phase 4 Study of Fluid Infusion During Breast Surgery.
Brief Title: Fluid Infusion During Breast Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Mastectomy opti.
Record Dates: First submitted 2007-02-05; First posted 2007-02-06 (Estimated); Last update posted 2009-03-03 (Estimated); Status verified 2009-02

CONDITIONS: Breast Surgery
Keywords: Fluid Therapy; Crystalloid; Colloid; Perioperative; Optimization; Goal-directed Therapy
MeSH Terms: interventions — Ringer's Lactate

INTERVENTIONS:
Drug: Hydroxyethylstarch 130/0,4
Drug: Lactated Ringer's solution

SUMMARY:
The investigators want to investigate the effects of two different kinds of fluid infusions given during varicose vein surgery. Both types of fluid are regularly given during surgery, and the investigators want to compare their respective effects on balance, nausea/vomiting and orthostatic function after surgery.

The investigators' hypothesis is that using a colloid solution will improve orthostatic function, balance, nausea/vomiting and reduce hospital stay.

DETAILED DESCRIPTION:
The optimal amount and type of fluid given during surgery has not been defined. It has been agreed that hypovolemia must be avoided, but at the same time it has been agreed that fluid excess is harmful for organ function.When distributing fluids it is usually either crystalloids og colloids which are given. The effects of the two types of fluid have not been compared. Our hypothesis is that using a colloid (HES 130/0,4) will improve orthostatic function, nausea/vomiting and shorten hospital stay, compared to using a crystalloid (Lactated Ringer's solution).The amount of fluid the patient receives, will be individually tailored by monitoring SV using esophageal Doppler technique during surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients having performed elective breast surgery.
* Age between 18 and 70 years
* Patients who have given written consent to participate in the project after haven completely understood the contents and limitations of the protocol.

Exclusion Criteria:

* Patients who do not understand or speak Danish
* Patients who have not signed the informed consent or the written authority
* pre-medication, except 1g paracetamol
* ASA > II
* Pregnant or breastfeeding
* Known to have Renal disease
* Known to have Psychiatric disorder (not considering the use of SSRI antidepressive)
* Need for crash induction or prone position.
* Oesophageal varicoses
* Necrosis or cancer in: Mouth, Pharynx, Larynx or Oesophagus
* Coarctation or aneurism in the proximal Aorta
* Severe bleeding disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2009-04; Primary Completion 2009-09 (Estimated); Study Completion 2009-09 (Estimated)

PRIMARY OUTCOMES:
To investigate orthostatic function, measured by Finapress

SECONDARY OUTCOMES:
To investigate the occurrence of postsurgery nausea/vomiting.
To investigate the amount of time until discharge criteria from the Postanaesthetic Care Unit have been achieved.
To investigate balance function, measured by BalanceMaster

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Kehlet, M.D. Ph.d., Study Director — dept of surgical patophysiology
Locations (1):
- Dept of anesthesia 2041, ABD centre, Rigshospitalet, Blegdamsvej, Copenhagen, Region Sjælland, Denmark